CLINICAL TRIAL: NCT06861881
Title: Continuous Glucose Monitoring in Patients Undergoing Cardiopulmonary Bypass
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00125789
Record Dates: First submitted 2025-02-20; First posted 2025-03-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus)
Keywords: continuous glucose monitoring; cardiopulmonary bypass; cardiac surgery
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continuous Glucose Monitoring (Experimental): All participants will wear the Dexcom G7 continuous glucose monitor continuously during their cardiothoracic surgery and throughout their time admitted to the Cardiovascular Intensive Care Unit.
  Interventions: Device: Dexcom G7 Continuous Glucose Monitor

INTERVENTIONS:
Device: Dexcom G7 Continuous Glucose Monitor — Dexcom G7 continuous glucose monitor will be placed prior to cardiac surgery. It will be worn continuously throughout the perioperative period and during the time admitted to the Cardiovascular Intensive Care Unit.

SUMMARY:
The purpose of this research study is to test the accuracy of the Dexcom continuous glucose monitoring device during the cardiothoracic surgical procedure and recovery period in the Cardiac Intensive Care Unit. Readings from the device will be compared with the standard of care blood glucose levels that are obtained during your surgery and postoperatively.

DETAILED DESCRIPTION:
The proposed study would examine 100 adult patients specifically undergoing cardiac surgical procedures with the explicit goal of comparing continuous glucose monitoring accuracy to point-of-care testing, particularly in the setting of physiologic perturbations due to vasopressors, acidosis, and hypothermia. With a large sample size and few stipulations on the included patients, this well-powered study would give broadly applicable guidance regarding continuous glucose monitoring use in this population. The study would establish a pathway to further research regarding optimizing continuous glucose monitoring accuracy, providing earlier detection of out-of-range glucose values, improving the precision of insulin titration, and ultimately improving glucose control in the cardiac surgical population, which may improve patient outcomes, including mortality. This would be the first study to describe intraoperative use of the newest Dexcom continuous glucose monitoring device, the G7, which has the shortest available warmup time and may be the most accurate continuous glucose monitoring device on the market.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing cardiac surgery with cardiopulmonary bypass at Atrium Health Wake Forest Baptist Medical Center

Exclusion criteria:

* Under 18 years of age
* Pregnant women
* Patients with a contraindication to device placement on the posterior arm, including rash, missing extremity, or existing line or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Continuous Glucose Monitoring Accuracy Compared to Point-of-Care Measurements | Up to Day 10
  Glucose values (mg/dL) from the continuous glucose monitoring will be compared to glucose values obtained from point-of-care arterial blood gas and/or fingerstick capillary glucose measurements.
Percentage of Continuous Glucose Monitoring Accuracy with Vasopressor Use | Up to Day 10
  Glucose values from the continuous glucose monitoring will be compared to glucose values obtained from point-of-care arterial blood gas measurements when vasopressors are utilized for hemodynamic optimization.
Percentage of Continuous Glucose Monitoring Accuracy with Hypothermia | Day 1
  Glucose values from the continuous glucose monitoring will be compared to glucose values obtained from point-of-care arterial blood gas measurements during the hypothermic period intraoperatively.
Percentage of Continuous Glucose Monitoring Accuracy with Acidosis | Up to Day 10
  Glucose values from the continuous glucose monitoring will be compared to glucose values obtained from point-of-care arterial blood gas measurements intraoperatively when the participant is acidotic.

SECONDARY OUTCOMES:
Incidence of Continuous Glucose Monitor Malfunction | Up to Day 10
  Number of times the Dexcom G7 continuous glucose monitor malfunctioned during use, including sensor loss or monitor failure.
Duration of Time Continuous Glucose Monitor Experienced Sensor Loss | Up to Day 10
  Amount of time the Dexcom G7 continuous glucose monitor experienced sensor loss while in use.
Continuous Glucose Monitor Measurement Expenses | Up to Day 10
  Total expenditures to the patient for the costs of all glucose measurements (arterial blood gases, glucometers as point of care, laboratory drawn glucose measurements - included in metabolic profile laboratory measurements as well) obtained during the course of wearing the continuous glucose monitoring device compared to the cost of the Dexcom G7 continuous glucose monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Hicks, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No